CLINICAL TRIAL: NCT02378571
Title: Telemonitoring Adherence to Medications to Reduce Heart Failure Readmissions: A Pilot Randomized Clinical Trial
Brief Title: Medication Adherence Telemonitoring to Reduce Heart Failure Readmissions
Acronym: TEAM-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Principal Investigator, Ian Kronish, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAO3305
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure
Keywords: Medication adherence; Hospital readmissions
MeSH Terms: conditions — Heart Failure; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): Participants assigned to usual care will also be provided with a GlowCap prior to discharge and will be instructed to take their loop diuretic from this bottle and to notify the study team about prescribed dose changes. This information, however, will solely be used to measure medication adherence and will not be provided to a member of the study team nor to any of the participants' health care providers until the completion of the study period, at least 1 month later. Participants will not be provided with any advice on heart failure adherence.
- Medication adherence telemonitoring (Experimental): At discharge, participants in the intervention group will be instructed to take their loop diuretic exclusively from the GlowCap in the manner prescribed by their physician. A study team member will review the adherence data on a daily basis (except holidays and weekends) during the first 7 days after discharge, and then on, at minimum, a weekly basis. The study team member will respond to adherence data using clinical judgment as they would if the information was obtained during clinical care. Specifically, when contacting nonadherent participants, the member of the study team will provide participants with feedback on their electronic adherence; will inquire about potential consequences of missed doses; and will assess and respond to reasons for missed doses.
  Interventions: Behavioral: Medication adherence telemonitoring

INTERVENTIONS:
Behavioral: Medication adherence telemonitoring — The member of the study team will respond to adherence data using clinical judgment as they would if the information was obtained during clinical care. Specifically, when contacting nonadherent participants, the member of the study team will provide participants with feedback on their electronic adherence; will inquire about potential consequences of missed doses; and will assess and respond to reasons for missed doses.
  Arms: Medication adherence telemonitoring

SUMMARY:
The overall purpose of this project is to determine the feasibility of conducting a large scale randomized clinical trial that compares remote monitoring of adherence to loop diuretics using a wireless electronic pillcap with usual care among recently hospitalized heart failure patients. The long-term goal of this program of research is to determine the effect of the adherence telemonitoring intervention on medication adherence and hospital readmissions among recently hospitalized heart failure patients.

DETAILED DESCRIPTION:
Approximately one in four patients hospitalized with heart failure is readmitted within 30 days of discharge and more than 50% are readmitted within 6 months of discharge. Heart failure admissions are a major contributor to the enormous health care costs associated with heart failure. Thus far, the identification of effective interventions that prevent unnecessary readmissions has remained elusive. As a result, there is a pressing need to identify novel, cost-effective approaches to reducing heart failure readmissions. A growing body of research suggests that poor adherence to heart failure medications is a major reason for preventable heart failure readmissions. In particular, loop diuretic medications are essential to preventing the cardiopulmonary system from becoming overloaded. Patients who have been recently hospitalized may be especially vulnerable to adherence problems as a result of the stress of the recent hospitalization which commonly induces sleep deprivation, nutritional deficiency, physical deconditioning, cognitive impairment, and even delirium. Recent advances in wireless health now enable us to remotely, unobtrusively, and objectively monitor adherence to heart failure medications in the post-discharge period. Early identification of non-adherence to loop diuretic medications has the prevention to prevent a volume overloaded state that leads to a heart failure readmission. As patients who are non-adherent to their loop diuretics may also be non-adherent to other recommended self-management behaviors, early identification of medication nonadherence may provide the context to identify other gaps in self-management. To test our hypothesis that it is feasible to conduct a randomized trial of wireless, medication adherence monitoring with feedback to patients and clinicians, the investigators will enroll 40 patients who are hospitalized for heart failure and discharged on a diuretic medication. Patients will be randomized to 1) usual heart failure care + telemonitoring adherence to diuretic medications (INT); N=20 or 2) usual heart failure care (CTR); N=20. All patients will be asked to take their diuretic medication from a standard pill bottle covered by an electronic pill cap (GlowCap), but only patients assigned to the intervention arm will have their adherence telemonitored by a study clinician in real-time. Patients will have their adherence to medications measured in this fashion for 30 days after discharge. Patients will be contacted at 30 days to determine if they have been hospitalized and to collect other self-reported outcomes data.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for heart failure
* Prescribed loop diuretic medication at discharge

Exclusion Criteria:

* Age less than 21 years
* New York Heart Association Class IV heart failure
* Terminal illness (<6 mo prognosis)
* Unable to self-administer medications due to mental illness or cognitive impairment
* Non-English/Spanish speaking
* Discharged to an institutional setting (e.g., nursing home)
* Cardiologist or primary care provider refusal
* Unavailable for follow-up
* No access to telephone
* Enrolled in another cardiac trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percentage of days participants take the correct number of doses of their diuretic | 30 days post-discharge
  Loop diuretic adherence: Adherence to the diuretic medication will be electronically measured using GlowCaps (Vitality Inc.) in the 30 days after hospitalization. Medication adherence will be calculated as the percent of days participants take the correct number of doses of their diuretic. Days when participants are incapable of taking their medication from the GlowCap bottle (e.g., while hospitalized) will be censored from calculations.

SECONDARY OUTCOMES:
Score on the Self Care Heart Failure Index | 30 days post-discharge
  Heart Failure Symptoms, Self-Efficacy for self-managing heart failure, and Self-Management Behaviors will be measured using Self Care Heart Failure Index
Proportion very or extremely satisfied with heart failure care | 30 days post-discharge
  Satisfaction with Heart Failure Care will be assessed by asking participants "Overall, how satisfied are you with the care you have been receiving for your heart problems over the last 30 days?" Response options will include: "not at all satisfied", "a little satisfied", "very satisfied," and "extremely satisfied."
Number of readmissions and emergency room visits | 30 days post-discharge
  Readmissions and emergency room visits will be assessed by contacting participants or their close contacts at 30 days. Hospital records will be reviewed to confirm readmissions, to determine the reason for readmission or emergency room visit (heart failure versus other), and to determine whether it was related to medication nonadherence.
Proportion attending at least 1 scheduled outpatient clinic visit within 30 days of discharge | 30 days post-discharge
  Attendance at scheduled outpatient clinic visits will be assessed by contacting participants or their close contacts at 30 days. Hospital records will be reviewed, when available, to determine whether and how medication adherence was addressed during the visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Kronish, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Gallagher BD, Moise N, Haerizadeh M, Ye S, Medina V, Kronish IM. Telemonitoring Adherence to Medications in Heart Failure Patients (TEAM-HF): A Pilot Randomized Clinical Trial. J Card Fail. 2017 Apr;23(4):345-349. doi: 10.1016/j.cardfail.2016.11.001. Epub 2016 Nov 3. PMID 27818309